CLINICAL TRIAL: NCT03495882
Title: A Phase 1 / 2, Open-Label, Multi-Arm Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Biological, and Clinical Activity of AGEN1884 in Combination With AGEN2034 in Subjects With Metastatic or Locally Advanced Solid Tumors, and Expansion Into Select Solid Tumors
Brief Title: Subjects With Metastatic or Locally Advanced Solid Tumors, and Expansion Into Select Solid Tumors (Cervical)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-550-01
Record Dates: First submitted 2018-01-19; First posted 2018-04-12 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AGEN1884 + AGEN2034 (Experimental): AGEN1884 in combination with AGEN2034 in subjects with Subjects with Metastatic or Locally Advanced Solid Tumors, and Expansion into Select Solid Tumors (cervical)
  Interventions: Drug: AGEN1884 + AGEN2034

INTERVENTIONS:
Drug: AGEN1884 + AGEN2034 — AGEN1884 + AGEN2034 according to protocol design

SUMMARY:
This is a Phase 1/2, open-label study of AGEN1884 in combination with AGEN2034 in subjects with locally advanced, recurrent and/or metastatic solid tumors including cervical cancer. AGEN2034 is a novel, fully human monoclonal immunoglobulin G4 (IgG4) antibody, designed to block program cell death-1 (PD-1). AGEN1884 is a novel, fully human monoclonal immunoglobulin G1 (IgG1) antibody, designed to block cytotoxic T-lymphocyte antigen-4 (CTLA-4).

DETAILED DESCRIPTION:
The trial consists of 2 phases:

* Phase 1: Dose escalation
* Phase 2: Expansion in advanced cervical cancer

Phase 1: Dose Escalation:

The enrollment to the Phase 1 portion of the study is completed. The trial will consist of a 3+3 dose escalation that will evaluate different combination dose levels (CDL) of AGEN1884 and AGEN2034 in subjects with locally advanced, recurrent and/or metastatic solid tumors.

Subjects may be enrolled to the following CDL cohorts:

* CDL1 - AGEN1884 1 mg/kg every 6 weeks + AGEN2034 1 mg/kg every 2 weeks (starting CDL)
* CDL2 - AGEN1884 1 mg/kg every 6 weeks + AGEN2034 3 mg/kg every 2 weeks (maximum planned CDL)
* CDL-1 - AGEN1884 0.3 mg/kg every 6 weeks + AGEN2034 1 mg/kg every 2 weeks (potential de-escalation CDL)

Combination Dose Level 1 (CDL1) will be the first to be tested. Dose escalation will continue until the maximum planned CDL (CDL2) is shown to be safe or the maximum tolerated dose (MTD) is reached. The MTD is defined as the CDL below which ≥ 33% of subjects develop dose-limiting toxicities (DLT). The decision to escalate to the next cohort will be made by a Safety Monitoring Committee (SMC), based on safety assessments after all subjects of a cohort reached the end of the DLT observation period of 21 days. Should ≥2 DLTs be observed in CDL1, the SMC may open enrollment to CDL-1. The SMC will also select the CDL for Phase 2.

Each subject will receive the combination treatment for a maximum of 24 months or until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the trial or the investigational medicinal products (IMPs) occur. Subjects who do not complete the DLT observation period of 21 days after the first dose, for reasons other than a DLT will be replaced. Additional subjects will be backfilled, concurrently with the 3+3 dose escalation schema at the lower cleared CDL, to ensure that each cohort enrolls at least 10 subjects. These additional subjects at each dose level will have the purpose of generating additional safety, PK, and receptor occupancy (RO) data, and will not undergo formal DLT observation.

The SMC selected CDL2 (AGEN1884 1 mg/kg every 6 weeks + AGEN2034 3 mg/kg every 2 weeks) as the Recommended Phase 2 dose (RP2D).

Phase 2: Expansion in Select Tumors

To further characterize safety and efficacy, the following expansion cohort will be enrolled:

Advanced cervical cancer In Phase 2, the RP2D of AGEN2034 and AGEN1884 will be administered for a maximum of 2 years or until confirmed progression, unacceptable toxicity, or any criterion for stopping the study drugs or withdrawal from the trial occurs.

For the Phase 2 portion of the trial, an Independent Data Monitoring Committee (IDMC) will be established to evaluate safety and efficacy and an IERC will be established to adjudicate tumor response.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this trial the subject must:

1. Voluntarily agree to participate by giving written informed consent. (Participation in pharmacogenomics testing is optional.)
2. Be ≥18 years of age.
3. Diagnosis:

   1. Phase 1: Male or female having a histologically or cytologically confirmed diagnosis of a locally advanced, recurrent, and/or metastatic solid tumor for which no standard therapy is available or standard therapy has failed.
   2. Phase 2:

   I. Female having (1) a histologically or cytologically confirmed diagnosis of squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix, and (2) locally advanced, recurrent, and/or metastatic disease at the time of enrollment. Histologic confirmation of the original primary tumor is required via pathology report.

   Note: The following cervical tumors are not eligible: minimal deviation/adenoma malignum, gastric type adenocarcinoma, clear cell carcinoma, and mesonephric carcinoma.

   II. Has cervical cancer and has relapsed after a platinum-based treatment (first line) regimen for locally advanced, recurrent, and/or metastatic disease; Note: Subjects who only received platinum-based chemotherapy concurrently with primary radiation (e.g., weekly cisplatin) or adjuvant chemotherapy following completion of radiation therapy (e.g., paclitaxel and carboplatin for ≤4 cycles) and progressed within 6 months after treatment completion will be eligible as this systemic therapy will be considered first line.
4. Measurable Disease:

   1. Phase 1: Have objective evidence of disease; the presence of measurable disease is not required.
   2. Phase 2: Have measurable disease on imaging based on RECIST version 1.1. Note: Subjects must have at least one "target lesion" to be used to assess response, as defined by RECIST version 1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented, or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.

   Note: Measurable disease by RECIST 1.1 must be confirmed by independent central radiologic review prior to first dose. Subjects without centrally confirmed measurable disease at baseline will not be eligible for this trial.
5. Have a life expectancy of at least 3 months and an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Have adequate organ function as indicated by the following laboratory values:

   1. Adequate hematological function defined by absolute neutrophil count (ANC) ≥1.5 x 10^9/L, platelet count ≥100 x 10^9/L, and hemoglobin

      ≥8 g/dL (without transfusions within 1 week of first dose).
   2. Adequate hepatic function based on a total bilirubin level <1.5 x the institutional upper limit of normal (IULN), aspartate aminotransferase (AST) level ≤2.5 x IULN, alanine aminotransferase (ALT) level ≤2.5 x IULN, and alkaline phosphatase ≤2.5 IULN.
   3. Adequate renal function defined as creatinine ≤1.5 x IULN OR calculated creatinine clearance ≥50 mL/min for subjects with creatinine levels >1.5 x IULN (if no local guideline is available, creatinine clearance should be calculated using the Cockcroft-Gault Method).
   4. Adequate coagulation defined by international normalized ratio (INR) or prothrombin time ≤1.5 x IULN (unless the subject is receiving anticoagulant therapy); and activated partial thromboplastin time (aPTT) ≤1.5 x IULN (unless the subject is receiving anticoagulant therapy)
7. Other than the cancer for which the subject is enrolled, have no history of prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous-cell carcinoma of the skin, or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.

   Note: In Phase 2, the history and time requirement for no evidence of disease for 5 years does not apply to the cancer for which the subject is enrolled in the trial.
8. In Phase 2, subjects must provide a sufficient and adequate formalin fixed paraffin embedded (FFPE) tumor tissue sample preferably from the most recent biopsy of a tumor lesion, collected either at the time of or after the diagnosis of locally advanced, recurrent, and/or metastatic disease has been made AND from a site not previously irradiated. If no tumor tissue is available, a fresh biopsy will be required.

   Note: Tissue from needle or excisional biopsy or from resection is required.
9. Female subjects must have a negative serum pregnancy test at screening (within 72 hours of first dose of study drug) if of childbearing potential or be of non- childbearing potential. Non-childbearing potential is defined as (by other than medical reasons):

   1. ≥45 years of age and has not had menses for greater than 1 year,
   2. Amenorrheic for ≥ 2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone (FSH) value in the postmenopausal range upon pretrial (screening) evaluation,
   3. Whose status is post hysterectomy, oophorectomy, or tubal ligation.
10. If of childbearing potential, female subjects must be willing to use 2 highly effective contraceptive measures (defined in the informed consent form [ICF]) throughout the study, starting with the screening visit through 120 days after the last dose of study drug.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the subject.
11. Male subjects with a female partner(s) of childbearing potential must agree to use 2 highly effective contraceptive measures (defined in the ICF) throughout the trial starting with the screening visit through 120 days after the last dose of study drug is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the subject.
12. Is willing and able to comply with the requirements of the protocol.

Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving trial therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has an inadequate washout period prior to first dose of study drug defined as:

   1. Received systemic cytotoxic chemotherapy or biological therapy within 3 weeks before first dose,
   2. Received radiation therapy within 3 weeks before first dose, or
   3. Had major surgery within 4 weeks before first dose.
3. Has received prior therapy with:

   1. Any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints) such as anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibodies
   2. For Phase 2: >1 systemic treatment regimen for the locally advanced recurrent, and/or metastatic cervical cancer for which the subject is considered for the study. Subjects who received a systemic regimen immediately after progressing within 6 months of completing chemotherapy concurrent with primary radiation or adjuvant chemotherapy after radiation will only be considered as having 1 prior systemic regimen for the purpose of this criterion.

   Note: In Phase 1, prior treatment with a CTLA-4 antibody is permissible for subjects with metastatic melanoma.
4. Has persisting toxicity related to prior therapy of National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI-CTCAE) Grade >1 severity.

   Note: Sensory neuropathy or alopecia of Grade ≤2 is acceptable.
5. Is expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
6. Has known severe hypersensitivity reactions to fully human monoclonal antibodies (NCI-CTCAE Version 4.03 Grade ≥3), any history of anaphylaxis, or uncontrolled asthma.
7. Is receiving systemic corticosteroid therapy ≤7 days prior to first dose of study treatment or receiving any other form of systemic immunosuppressive medication (corticosteroid use on study for management of immune-related adverse events (AE), and/or a premedication for intravenous (IV) contrast allergies/reactions is allowed). Subjects who are receiving daily corticosteroid replacement therapy are an exception to this rule. Examples of permitted therapy are daily prednisone at doses of 5 to 7.5 mg or equivalent hydrocortisone dose, and steroid therapy administered by topical, intraocular, intranasal, and/or inhalation routes.
8. Has a central nervous system (CNS) tumor, metastasis(es), and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period OR identified prior to consent.

   Note: Subjects with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at screening (based on 2 sets of brain images performed ≥4 weeks apart, and obtained after the brain metastases treatment). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be minimal and be expected as sequelae from treated lesions. For individuals who received steroids as part of brain metastases treatment, steroids must be discontinued ≥7 days prior to first dose of study drug.
9. Has active or history of autoimmune disease that has required systemic treatment within 2 years of the start of study treatment (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of immunosuppressive systemic treatment.

   Note: Subjects with diabetes type 1, vitiligo, psoriasis, hypo-, or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
10. Has had an allogeneic tissue/solid organ transplant.
11. Has or had interstitial lung disease (ILD) OR has had a history of pneumonitis that has required oral or IV corticosteroids.
12. Has an active infection requiring IV systemic therapy.
13. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
14. Has known active Hepatitis B, Hepatitis C, or tuberculosis. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
15. Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥II), or serious uncontrolled cardiac arrhythmia requiring medication.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
19. Is legally incapacitated or has limited legal capacity.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of AGEN2034 and/or AGEN1884.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR), as determined by IERC, in the analysis population | Evaluated throughout the protocol, up to 2 years.
  per RECIST 1.1

SECONDARY OUTCOMES:
Safety and Tolerability of AGEN2034 and AGEN1884 | From the time of the first dose to the end of follow-up (up to 2 years after the last dose).
  Frequency, severity, and duration of TEAEs and laboratory abnormalities, using NCI CTCAE v4.03.
Maximum drug concentration observed postdose at steady-state (Cmax-ss) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Minimum observed concentration at steady-state (Cmin-ss) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Area under the drug concentration-time curve within time span t1 to t2 at steady-state (AUC(τ1-τ2)-ss) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Area under the drug concentration-time curve from time zero to time t (AUC(0-t)), area under the drug concentration-time curve from time zero to infinity (AUC(0-∞)) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Time to maximum observed concentration (tmax) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Terminal disposition rate constant (λz) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Terminal elimination half-life (t1/2) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Systemic clearance (CL) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Volume of distribution (Vd) | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Immunogenicity of AGEN2034 and AGEN1884 | Pre-dose through 3 months after last dose.
  Serum AGEN2034 and AGEN1884 ADA concentrations and serum AGEN2034 and AGEN1884 concentrations measured throughout the study.
Objective Response Rate (ORR), as determined by investigator | Evaluated throughout the protocol, up to 2 years.
  per RECIST 1.1
Duration of Response (DOR) | Time from first observation of response to first observation of documented disease progression, up to 3 years.
  per RECIST 1.1, as determined by an IERC and investigator, defined as time from first observation of response to first observation of documented disease progression (or death within 12 weeks after last tumor assessment). Subjects without an event at analysis cutoff date will be censored on date of last tumor assessment.
Disease Control Rate (DCR) | Duration of the trial, up to 3 years.
  defined as proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD) for at least 12 weeks.
Duration of Stable Disease (SD) | Duration of the trial, up to 3 years.
  measured from the start of treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including baseline measurements.
Time to Response | Duration of the treatment phase of the trial, up to 2 years.
  defined as the time from the first dose date to first observation of confirmed response.
Progression-free Survival (PFS) | Duration of the treatment phase of the trial, up to 2 years.
  defined as time from first treatment administration to first observation of documented disease progression (or death within 12 weeks after last tumor assessment), per RECIST 1.1, as determined by an IERC and investigator. Subjects without an event at analysis cutoff date will be censored on date of last tumor assessment.
Overall Survival Rate (OS) | Duration of the treatment phase of the trial, up to 2 years.
  defined as time from start of treatment to death. For subjects who are still alive at time of data cutoff for trial analysis or who are lost to follow-up, survival will be censored at the last recorded date that the subject is known to be alive as of the cutoff date for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (47):
- United States (13):
  - Comprehensive Care and Research Center, Goodyear, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of Miami, Miami, Florida
  - BRCR Medical Center, Inc, Plantation, Florida
  - Augusta University, Augusta, Georgia
  - Cancer Treatment Centers of America, Zion, Illinois
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Chattanooga's Program In Women's Oncology, Chattanooga, Tennessee
  - CliniCore International, Baytown, Texas
  - Providence Regional Cancer System, Aberdeen, Washington
  - Swedish Cancer Institute, Seattle, Washington
- Australia (4):
  - Linear Clinical Research, Perth, Western Australia
  - Mater Research, South Brisbane
  - Icon Cancer Care South Brisbane, South Brisbane
  - Scientia Clinical Research, Sydney
- Brazil (2):
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda., São Paulo
  - IBCC - Instituto Brasileiro de Controle do Câncer, São Paulo
- LLC Arensia Exploratory Medicine, Tbilisi, Georgia
- Hungary (8):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem, Debrecen
  - Bacs-Kiskun Megyei Korhaz, Kecskemét
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- ARENSIA Exploratory Medicine Unit, Institute of Oncology, Chisinau, Moldova
- Poland (2):
  - BioResearch Group SP. Z O.O., Nadarzyn
  - Centrum Onkologii-Instytut im.M.Sklodowskiej Curie, Warsaw
- Spain (6):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - START Madrid. Oncology Phase I, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Ukraine (10):
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipro
  - CI Transcarpathian Cl Onc Center Dep of Surgery #1 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
  - CI of Healthcare Regional Clinical Specialized Dispensary of the Radiation Protection, Department of Surgery, Kharkiv
  - Khmelnytskyi Regional Oncological Dispensary, Khmelnytskyi
  - Medical Clinic Innovacia, LLC, Kiev
  - Kyiv Сity Clinical Oncological Center, Kyiv
  - Medical Center Oncolife, Kyiv
  - Limited Liability Company Company Adonis, Kyiv
  - Treatment-Prevention Institution Volyn Regional Oncological Dispensary, Lutsk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Malley DM, Neffa M, Monk BJ, Melkadze T, Huang M, Kryzhanivska A, Bulat I, Meniawy TM, Bagameri A, Wang EW, Doger de Speville Uribe B, Hegg R, Ortuzar Feliu W, Ancukiewicz M, Lugowska I. Dual PD-1 and CTLA-4 Checkpoint Blockade Using Balstilimab and Zalifrelimab Combination as Second-Line Treatment for Advanced Cervical Cancer: An Open-Label Phase II Study. J Clin Oncol. 2022 Mar 1;40(7):762-771. doi: 10.1200/JCO.21.02067. Epub 2021 Dec 21. PMID 34932394